CLINICAL TRIAL: NCT04868370
Title: Validation of a Novel Instrument Task for Assessing Upper Limb Sensorimotor Impairments in Persons With Chronic Neurological Disorders
Brief Title: Validation of a Novel Instrument Task for Assessing Upper Limb
Status: Completed | Type: Observational
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Kliniken Valens, Rehazentrum Valens, Taminaplatz 1, 7317 Valens (Unknown)
Responsible Party: Sponsor
Other Study IDs: BASEC 2021-00633
Record Dates: First submitted 2021-04-26; First posted 2021-04-30 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Assessment of Arm and Hand Sensorimotor Functions in Multiple Sclerosis Subjects
Keywords: Rehabilitation; Multiple Sclerosis; Sensorimotor Impairment; Assessments; Neurological Disease
MeSH Terms: conditions — Multiple Sclerosis; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis (MS)
  Interventions: Other: Assessment of the upper limb (VPIT + PPIT)
- Healthy Subject

INTERVENTIONS:
Other: Assessment of the upper limb (VPIT + PPIT) — Assessment of the upper limb sensorimotor function (VPIT and PPIT)
  Groups: Multiple Sclerosis (MS)

SUMMARY:
The aim of this study i to investigate a new approach (Physical Peg Insertion Test, PPIT) to measure sensorimotor function in the arm and hand. To achieve this, this novel approach will be compared with an existing approach (Virtual Peg Insertion Test, VPIT).

DETAILED DESCRIPTION:
In movement disorders, such as multiple sclerosis, impairments in sensorimotor control of goal-directed upper limb movements are commonly present, leading to a decreased ability to perform daily life activities and increased dependence on caregivers . Due to the disabling nature of upper limb impairments, they are often a focus during the neurorehabilitation process of persons with movement disorders. This process relies on a precise description of the presence and severity of sensorimotor impairments through so-called assessments. Specifically, these assessments are essential to individualize therapeutic interventions, to provide documentation for insurances justifying further therapy, and to shed light on the often unknown mechanisms underlying the impairments and their temporal evolution.

Technology-aided assessments can provide detailed movement (kinematic) and grip force (kinetic) data that allows an objective and traceable description of upper limb behaviour. This offers the potential to sensitively characterize sensorimotor impairments and could help significantly reducing sample sizes required in resource-demanding clinical trials. Such technology-aided assessments typically consist of a robotic interface (e.g., exoskeleton or end-effector) that functions as a joystick and a virtual reality environment with a goal-directed manipulation task that is rendered on a 2D computer screen located next to the robotic interface. While these approaches are widely used for research purposes and showed promising results in detecting sensorimotor impairments, certain subjects were observed to have atypical movement patterns and high variability when repeatedly performing the assessment task (high intra-subject variability). These artifacts can results from unintuitive perception of depth on the 2D screen and missing visuomotor collocation, which can induce a bias in the outcome measures of the assessment and reduce the ability of the assessment to capture longitudinal changes (reliability and sensitivity). To overcome these challenges, assessment tasks relying on virtual collocated visuomotor feedback or immersive head mounted displays have been proposed. However, the virtual collocated visuomotor feedback still has its limitations, especially when subjects are supposed to interact with the virtual objects, such as in 3D object manipulation tasks that are typically used in clinical settings. In addition, head mounted display are expected to have limited clinical feasibility in persons that are naïve to technologies or have cognitive impairments.

The aim of this collaborative project between ETH Zurich (Prof. Dr. Gassert, Dr. Lambercy, Dr. Kanzler) and the Kliniken Valens (Dr. med. Dr. sc. nat. Roman Gonzenbach, Ramona Sylvester) is to validate the concept of assessing upper limb sensorimotor impairments with a robotic interface embedded in a novel physical 3D object manipulation task, the Physical Peg Insertion Test (PPIT), and compare it to an existing virtual assessment approach. In more details, the aim is to perform a longitudinal study with the PPIT and its previously validated virtual pendent, the Virtual Peg Insertion Test (VPIT), in persons with movement disorders. This will allow to compare the feasibility, validity, reliability, and sensitivity of both physical and virtual instrumented assessments. Both approaches rely on a CE-certified haptic end-effector device (Geomagic Touch, 3D Systems) and an instrumented handle. For the PPIT, an electromagnet that can be controlled through the applied grip forces is attached to the end-effector and is required to pick up physical magnetic pegs in a physical pegboard task. For the VPIT, a personal computer renders a virtual reality environment with virtual pegs that need to be transported into virtual holes. These approaches have been developed at the Rehabilitation Engineering Laboratory of ETH Zurich and have been shown to be feasible, safe, and time-efficient (5 repetitions of the task, approximately 15 min duration per body side) in able-bodied controls, and persons with stroke, multiple sclerosis, or cerebellar ataxia that have mild to moderate disability levels. While the PPIT has only been developed rather recently, the VPIT has already been extensively used in clinical studies world-wide. Most importantly, the VPIT has already been successfully established as a clinical routine assessment for all persons with multiple sclerosis that are admitted to the Kliniken Valens and is therefore well known to the clinic, which provides the basis for the smooth implementation of the planned project. Through these and other previous tests, sensor data from 120 able-bodied subjects, that serve as a normative database, and over 200 persons with movement disorders could already be recorded. The collected raw kinematic and kinetic data is typically transformed through a signal processing framework into 10 sensor-based metrics that provide information on different aspects of task performance, including for example movement smoothness, accuracy, and speed. Given that the PPIT provides the same sensor data as the VPIT, the signal processing framework of the VPIT can also be applied to the data collected with the PPIT, allowing to extract the 10 sensor-based metrics in both scenarios and serves as a basis for their comparison.

ELIGIBILITY:
Cohort Group: Multiple Sclerosis

Inclusion Criteria:

* 18 years old
* mild to moderate upper lim disability
* no strong cognitive deficits
* no concomitant disease that might affect upper limb performance
* able to follow procedures and to give informed consent

Cohort Group: Healthy Subjects

Inclusion Criteria:

* 18 years old
* no cognitive deficits
* no concomitant disease that might affect upper limb performance and
* able to follow procedures and to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Impaired subjects, that suffer from Multiple Sclerosis must be 18 years old and have mild to moderate upper limb disability. Further, they have no strong cognitive deficits or concomitant disease that might affect upper limb performance and they must be able to follow procedures and to give informed consent.
  Healthy subjects must be 18 years old and must not have any concomitant disease that might affect upper limb performance. Further, they have no strong cognitive deficits and must be able to follow procedures and to give informed consent.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Validation of the Physical Peg Insertion Test (PPIT) | 2 years
  Validate the concept of assessing upper limb sensorimotor impairments with a physical, instrumented 3D object manipulation task (PPIT) by comparing the intra-subject variability, validity, reliability, and sensitivity of the approach to the one of an established, virtual instrumented 3D object manipulation task (VPIT).
Feasibility of the Physical Peg Insertion Test (PPIT) | 2 years
  To judge the feasibility, subjects will be asked to complete a standardized questionnaire based on the System Usability Scale. Subsequently, the 10 sensor-based metrics will be calculated for each assessment based on the same data processing pipeline.
Reliability of the Physical Peg Insertion Test (PPIT) | 2 years
  For describing reliability, the following analysis will be performed across multiple repetitions of the tasks at the same measurement timepoint: the systematic change (learning effects), the standard deviation (intra-subject variability), the intra-class correlation coefficients (ICC, ability to discriminate subjects), and the minimal detectable change (MDC, signal to noise ratio) will be calculated.
Sensitivity of the Physical Peg Insertion Test (PPIT) | 2 years
  The sensitivity of the assessment will be determined based on the number of subjects that the assessment indicates as having meaningful changes in sensorimotor function across the intervention. For this purpose, the magnitude of longitudinal changes will be compared to the noise level of the assessment, as defined by the MDC.
Validity of the Physical Peg Insertion Test (PPIT) | 2 years
  For describing discriminant validity, a receiver operating curve (ROC) analysis between able-bodied controls and persons with movement disorders will be performed to judge the ability of the metrics to detect sensorimotor impairments. For describing concurrent validity, the outcome measures from the PPIT and VPIT will be correlated (Person correlation coefficients) to conventional clinical scales of sensorimotor impairments (e.g., the Nine Hole Peg Test and Box and Block Test).

CONTACTS AND LOCATIONS:
Overall Officials: Roman R. Gonzenbach, MD, Principal Investigator — Rehazentrum Valens, Taminaplatz 1, 7317 Valens
Locations (1):
- Rehazentrum Valens, Valens, Canton of St. Gallen, Switzerland